CLINICAL TRIAL: NCT05319535
Title: Implementing a Caregiver Skills Training Program (Caregivers FIRST): Function QUERI 2.0 (QUE 20-023)
Brief Title: Implementing a Skills-Based Caregiver Training Program (Caregivers FIRST): Function QUERI 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 21-002
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Function; Functional Status
Keywords: Caregivers; Veterans; Training Programs; Informal Care; Implementation Science; Functional Independence

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomized trial (parallel-CRT): used in pragmatic evaluations of health program or policy interventions, where half the clusters (in this case, VA medical centers) are randomly assigned to two interventions: Foundational REP (active comparator) vs. Enhanced REP (experimental).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foundational REP (Active Comparator): Foundational REP uses the Replicating Effective Program implementation strategy and includes 5 elements that were developed and tested in the investigators' prior Function QUERI work: Stakeholder engagement; Toolkit; SharePoint access for clinical program training materials; Data dashboard to assist sites with tracking their own data; and Diffusion Networks to promote peer-to-peer sharing and implementation support.
  Interventions: Other: Implementation Strategy: Foundational REP
- Enhanced REP (Experimental): Enhanced REP begins with the same activities as Foundational REP. Sites randomized to receive Enhanced REP will continue with Foundational REP and also receive higher intensity support for a period of approximately 4 months. The higher intensity support will consist of facilitation, a process of interactive problem solving and support that occurs in a context of a supportive interpersonal relationship and CONNECT, a complexity science-based bundle of interaction-oriented activities designed to supplement implementation efforts by promoting team function and readiness for change. Facilitation will be provided by Function QUERI team members.
  Interventions: Other: Implementation Strategy: Enhanced REP

INTERVENTIONS:
Other: Implementation Strategy: Foundational REP — Among Caregivers FIRST sites that do not meet implementation adoption benchmarks, the goal is to test implementation intensification approaches, specifically Foundational REP vs. Enhanced REP. The investigators propose that low intensity implementation support that promotes adapting Caregivers FIRST for context and provides tools for ongoing Caregivers FIRST evaluation (defined as foundational REP), will be sufficient for some but not all sites to successfully incorporate Caregivers FIRST into routine practice.
  Arms: Foundational REP
Other: Implementation Strategy: Enhanced REP — Among Caregivers FIRST sites that do not meet implementation adoption benchmarks, the goal is to test implementation intensification approaches, specifically Foundational REP vs. Enhanced REP. The investigators posit that higher intensity strategies (defined as Enhanced REP) that directly influence teams' capacity and skills to effectively self-organize and problem-solve will lead to higher implementation adoption, penetration, fidelity, and value.
  Arms: Enhanced REP

SUMMARY:
Implementing a Skills-Based Caregiver Training (Caregivers FIRST): Function QUERI 2.0 aims to compare implementation strategies for large-scale spread of Caregivers FIRST, a group training for friend or family caregivers of Veterans. The goal is to use a type III effectiveness-implementation hybrid design framework to compare continuation of implementation strategies for 24 sites that do not meet implementation adoption benchmarks.

DETAILED DESCRIPTION:
Background/Purpose. Over 5 million former or current military personnel receive informal care in the home from family members or friends. Unintended impacts on caregivers can include strain, burden, burnout, and depression. Additionally, half of caregivers of Veterans with functional/cognitive limitations report unmet needs for training.

Caregivers FIRST (Caregivers Finding Important Resources, Support, and Training) is an evidence-based skills training program for caregivers of Veterans with cognitive and/or functional limitations. Caregivers FIRST promotes Veteran function and independence through caregiver skill training and support in a series of 4 proactive group classes to help general caregivers build self-care and psychological coping, health system navigation, and hands-on clinical skills.

As part of Implementing a Skills-Based Caregiver Training (Caregivers FIRST), the investigators plan to implement the Caregivers FIRST clinical program nationally in partnership with the VA Caregiver Support Program (maximum 150 VA medical centers). The investigators then plan to use a type III effectiveness-implementation hybrid design framework with 24 sites that do not meet implementation adoption benchmarks. Those enrolled sites will be randomized to receive standard implementation support (foundational Replicating Effective Programs or REP) or a higher-intensity implementation support (enhanced REP including additional facilitation, self-organization, and team building support). The investigators will compare continuation of foundational REP versus addition of higher intensity strategies.

Key questions: What VA Central Office and regional (VISN) partnerships and activities will enhance national dissemination of Caregivers FIRST? How should Caregivers FIRST clinical program be adapted to leverage site-specific resources and optimize sustainability? Are there differences in implementation outcomes (penetration, fidelity) at 6, 12, or 18 months between arms? What is the impact on effectiveness outcomes/quality metrics (quality of VA General Caregiver Program, Veteran days in the community) at implementing sites? How do sites experience implementation strategies in each arm? The investigators also plan to conduct an explanatory sequential mixed method design that includes qualitative data collection and analysis that will not be reported here.

Methodology. To evaluate implementation, the investigators will randomize sites (n=24) 1:1 to either foundational REP or enhanced REP. The investigators will use generalized linear models to examine the effect of foundational vs. enhanced REP on implementation outcomes at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Site inclusion criteria includes sites not meeting benchmarks for adoption of Caregivers FIRST and submission of a signed participation agreement.
* Enrolled sites will all be exposed to Foundational REP.
* Half of sites will be randomized to receive higher-intensity implementation support (Enhanced REP).

Exclusion Criteria:

* The eight Caregivers FIRST (formerly called iHI-FIVES) sites that have previously participated in Function QUERI (ClinicalTrials.gov Identifier: NCT03474380) will be excluded from enrollment in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney H Van Houtven, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Kelli D. Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Susan N. Hastings, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset may be created upon request. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format.
  Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication.
  No data or statistical code that could lead to re-identification of individuals will be released.
  Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form.
  Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset.
Time Frame: Available upon request.
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.

REFERENCES:
- [Derived] Hughes JM, Makaroun LK, Decosimo K, Tucker M, Dadolf J, Drake C, Zullig LL, Coffman CJ, Kota S, Sperber NR, Christensen L, Chadduck T, Allen KD, Hastings SN, Van Houtven CH. Development and Delivery of Enhanced Implementation Support to Disseminate a National Caregiver Skills Training Program. Innov Aging. 2024 Dec 17;9(1):igae107. doi: 10.1093/geroni/igae107. eCollection 2025. PMID 39872410
- [Derived] Decosimo K, Drake C, Coffman CJ, Sperber NR, Tucker M, Hughes JM, Zullig LL, Chadduck T, Christensen L, Kaufman B, Allen KD, Hastings SN, Van Houtven CH. Implementation intensification to disseminate a skills-based caregiver training program: protocol for a type III effectiveness-implementation hybrid trial. Implement Sci Commun. 2023 Aug 16;4(1):97. doi: 10.1186/s43058-023-00475-7. PMID 37587517
- [Derived] Hughes JM, Zullig LL, Choate AL, Decosimo KP, Wang V, Van Houtven CH, Allen KD, Nicole Hastings S. Intensification of Implementation Strategies: Developing a Model of Foundational and Enhanced Implementation Approaches to Support National Adoption and Scale-up. Gerontologist. 2023 Mar 21;63(3):604-613. doi: 10.1093/geront/gnac130. PMID 36029028

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Protocol Enrollment reflect the number of VA Facilities (sites) enrolled.
Units Other Than Participants: VA Facilities
Period: Overall Study
Arm/Group | Foundational REP | Enhanced REP
Started | NA; 12 VA Facilities (Primary and secondary outcomes were site level; therefore, the unit of analysis for this study was VA Facilities (sites).) | NA; 13 VA Facilities (Primary and secondary outcomes were site level; therefore, the unit of analysis for this study was VA Facilities (sites).)
Completed | NA; 12 VA Facilities (Primary and secondary outcomes were site level; therefore, the unit of analysis for this study was VA Facilities (sites).) | NA; 13 VA Facilities (Primary and secondary outcomes were site level; therefore, the unit of analysis for this study was VA Facilities (sites).)
Not Completed | NA; 0 VA Facilities | NA; 0 VA Facilities

BASELINE CHARACTERISTICS:
Population: Primary and secondary outcomes were site level; therefore, the unit of analysis for this study was VA Facilities (sites). Since outcome data was collected at the site level, these characteristics are not relevant and were not collected.
Units Other Than Participants: VA Facilities
Groups:
- Total: Total of all reporting groups
Arm/Group | Foundational REP | Enhanced REP | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (VA Facilities) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data was collected at the site level and these characteristics were not relevant and not collected.
  years
    number analyzed (VA Facilities) | 0 | 0 | 0
Sex: Female, Male [Count of Units; unit: VA Facilities] — Population: Data was collected at the site level and these characteristics were not relevant and not collected.
  VA Facilities
    Female | NA — Since data was collected at the site level, these characteristics are not relevant and were not collected. | NA — Since data was collected at the site level, these characteristics are not relevant and were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Since data was collected at the site level, these characteristics are not relevant and were not collected. | NA — Since data was collected at the site level, these characteristics are not relevant and were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Units; unit: VA Facilities] | NA — Unit of analysis for this study was VA Facilities. | NA — Unit of analysis for this study was VA Facilities. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: VA Facilities]
  United States | 12 | 13 | 25
Sites with prior implementation of Caregivers FIRST [Count of Units; unit: VA Facilities] — Models included the arm indicator variable in addition to the stratification variables used in randomization including prior implementation of Caregivers FIRST before study start (yes vs. no)).
  VA Facilities | 7 | 7 | 14
Low facility complexity [Count of Units; unit: VA Facilities] — Models included the arm indicator variable in addition to the stratification variables used in randomization include site complexity level (high complexity '1a', '1b' or '1c' vs. all others).
  VA Facilities | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Penetration 1
Description: Penetration is defined as the 1) percentage of caregivers who received consults for VA caregiver education and training services who attended at least one class.
Time Frame: 12 months (cumulative)
Population: Unit of analysis for this study was VA Facilities (site level); therefore, the Overall Number of Participants Analyzed is not available.
Measure: Mean (Standard Deviation); unit: percentage of caregivers
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 12 | 13
percentage of caregivers | 6.1 (4.5) | 8.3 (4.5)
Statistical Analysis 1: Comparison: Foundational REP vs Enhanced REP; Models included the arm indicator variable in addition to the stratification variables used in randomization (site complexity level (high complexity '1a', '1b' or '1c' vs. all others); prior implementation of Caregivers First (yes vs. no)); Test type: Superiority; p = 0.26, Regression, Linear; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-1.8 to 6.1]

2. Primary Outcome: Penetration 2
Description: Penetration is defined as the 2) number of classes delivered by site.
Time Frame: 12 months (cumulative)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of classes
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 12 | 13
number of classes | 5.5 (4.9) | 8.4 (5.6)
Statistical Analysis 1: Comparison: Foundational REP vs Enhanced REP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.11, negative binomial regression; rate ratio = 1.7, 95% CI 2-sided [0.9 to 3.4]

3. Secondary Outcome: Fidelity 1
Description: Fidelity will be measured by 1) the percentage of number of recommended classes delivered by site.
Time Frame: 12 months (cumulative)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of classes
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 12 | 13
percentage of classes | 68.8 (61.4) | 104.8 (70.3)
Statistical Analysis 1: Comparison: Foundational REP vs Enhanced REP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.17, Regression, Linear; Mean Difference (Final Values) = 37.6, 95% CI 2-sided [-18.1 to 93.3]

4. Secondary Outcome: Fidelity 2
Description: Fidelity will be measured by 2) number of caregivers attended at least one class by site.
Time Frame: 12 months (cumulative)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of caregivers
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 12 | 13
number of caregivers | 1.9 (1.0) | 2.4 (0.7)
Statistical Analysis 1: Comparison: Foundational REP vs Enhanced REP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.10, Regression, Linear; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.1 to 1.4]

5. Secondary Outcome: Fidelity 3
Description: Fidelity will be measured by 3) mean number of classes attended per caregiver.
Time Frame: 12 months (cumulative)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: classes attended per caregiver
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 12 | 13
classes attended per caregiver | 11.3 (8.8) | 13.2 (8.6)
Statistical Analysis 1: Comparison: Foundational REP vs Enhanced REP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.36, negative binomial regression; rate ratio = 1.3, 95% CI 2-sided [0.7 to 2.3]

6. Secondary Outcome: Adoption
Description: Adoption is defined as the number of VA Facilities meeting a threshold of four or more training classes delivered to a minimum of five caregivers.
Time Frame: 12 months (cumulative)
Population: as for outcome 1
Measure: Number; unit: VA Facilities
Units Other Than Participants: VA Facilities
Arm/Group | Foundational REP | Enhanced REP
Number analyzed (Participants) | NA | NA
Number analyzed (VA Facilities) | 12 | 13
VA Facilities | 6 | 10
Statistical Analysis 1: Comparison: Foundational REP vs Enhanced REP; Model included the arm indicator variable; Test type: Superiority; p = 0.17, Regression, Logistic; Odds Ratio (OR) = 3.3, 95% CI 2-sided [0.6 to 18.5]

ADVERSE EVENTS:
Description: Outcomes were site level; therefore, the unit of analysis for this study was VA Facilities (sites). All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for Veterans, caregivers or providers or at the site level.
Arm/Group | Foundational REP | Enhanced REP
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT05319535/Prot_SAP_000.pdf